CLINICAL TRIAL: NCT06487806
Title: SmokefreeSGM Español Pilot, Beta Testing a Text-based Smoking Cessation Intervention for Sexual and Gender Minority Groups Preferring Spanish Language
Brief Title: SmokefreeSGM Español Pilot, Beta Testing a Text-based Smoking Cessation Intervention for Sexual and Gender Minority(SGM) Groups Preferring Spanish Language
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: We are hiring staff
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Irene Tami-Maury, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-23-1004
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation
Keywords: lesbian, gay, bisexual, transgender, queer/questioning (one's sexual or gender identity), and intersex(LGBTQI)
MeSH Terms: conditions — Smoking Cessation; Homosexuality, Female; Homosexuality; Bisexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Beta testing group (Experimental)
  Interventions: Behavioral: SmokefreeSGM

INTERVENTIONS:
Behavioral: SmokefreeSGM — Participants will be asked to set a quit date within the next 15 days before being enrolled in the SmokefreeSGM Español text messaging program. They will be mailed a 6-week supply of nicotine patches. The participants will get daily text messages for 6 weeks that will encourage them to quit smoking.

SUMMARY:
The purpose of this study is to test the usability, engagement and acceptability of SmokefreeSGM Español, a culturally and linguistically tailored version of SmokefreeSGM, among Spanish-speaking SGM smokers.

ELIGIBILITY:
Inclusion Criteria:

* Currently live in the United States
* Have smoked at least 100 cigarettes in their lifetime, smoke every day, and smoke ≥ 5 cigarettes a day
* Are willing to quit smoking in the next 15 days
* Have a cell phone number with an unlimited short message service (SMS) plan
* Have a positive cotinine saliva test to indicate their smoking status
* Speak fluent Spanish

Exclusion Criteria:

* Have a prepaid cell phone plan (pay-as-you-go plan)
* Have a cell phone number that does not work and/or is registered to someone else
* Have inadequate equipment/devices (i.e., webcam, speakers, mic) for participating in telehealth sessions via Microsoft Teams, Webex, or Zoom AND cannot meet in-person
* Pregnant or breastfeeding persons (nicotine patches are not generally recommended to this groups since nicotine can affect fetal and neonatal brain development)
* Contraindication for nicotine patches. Absolute contraindications include: severe eczema or serious skin conditions, allergy to nicotine patches, pregnancy, breastfeeding, heart attack in the past 2 months, ongoing angina, peptic ulcer disease, arrhythmia, or uncontrolled blood pressure. Potential contraindications include: stroke in the past 6 months, insulin therapy, and a current diagnosis of liver, kidney, or heart disease. Study participants reporting a potential contraindication will require approval from their primary care provider and/or other treating physician (e.g., psychiatrist) to use nicotine patches. If the request is denied or not returned in 2 weeks, potential study participants will be excluded from the study.
* Current use of tobacco cessation medications
* Current use of tobacco products other than cigarettes or electronic nicotine delivery systems (ENDS) (i.e., (e.g., cigar, cigarillo, little cigar, pipe, Hookah)
* Enrollment in another smoking cessation study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as an LGBTQ+ individual
Enrollment: 20 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Perceived Usability as Assessed by the System Usability Scale (SUS) | end of intervention (1month after quit date)
  This is a 10-item questionnaire. Total score ranges from 0 to 100, with a higher score indicating greater usability and a score above 75 indicating better outcome
Engagement with the text-messaging program as assessed by number of text messages a participant sends, including replies to the bidirectional texts messages of SmokefreeSGM Español program | end of intervention (1month after quit date)
Acceptability at 1 month as Assessed by the System Usability Scale (SUS) | end of intervention (1month after quit date)
  This is a 10-item questionnaire. Total score ranges from 0 to 100, with a higher score indicating greater acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Irene Tami-Maury, DMD, MSc, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No